CLINICAL TRIAL: NCT06407570
Title: Dysphagia and Quality of Life in Patients With Oral Squamous Cell Carcinoma Before and After Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: CCOdysphagia
Record Dates: First submitted 2024-04-22; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Oral Cavity Cancer; Dysphagia; Quality of Life
Keywords: Oral Cavity Cancer; Dysphagia; Quality of Life; Days alive and out of hospital; Rehabilitation
MeSH Terms: conditions — Mouth Neoplasms; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While the group of oral cavity cancer (OCC) survivors continue to increase, surgeons and oncologist intensify their search for improved treatment and rehabilitation methods to reduce the morbidity of management without compromising the oncological safety. The predominant problem after treatment of OCC is dysphagia, which is associated with malnutrition, aspiration pneumonia, hospital re-admission, and reduced quality of life (QoL) and survival.

In a pilot study, the investigators found that 45% of OCC patients reported significant eating disabilities two years after surgical treatment. However, the international literature is limited on the dysphagia and QoL of OCC survivors.

With an overall goal to improve the QoL and health status in patients treated for OCC, the present study aims to

1. systematically evaluate the swallowing function before and after treatment,
2. investigate the impact of swallowing function on QoL,
3. identify risk factors for dysphagia,
4. investigate if swallowing function is an independent factor for the number of ´days alive and out of hospital´
5. evaluate the rehabilitation offered to OCC patients in Danish municipalities and the effect on swallowing outcomes.

One hundred patients treated for OCC will be included prospectively during a 2-year period. Data on type and location of tumour, treatment modality, complications, patient weight, dietary intake, rehabilitation program, hospital admissions, recurrences, and survival will be collected. Questionnaires and Modified Barium Swallow Study (MBSS) will be performed before and 2 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma with any location in the oral cavity including recurrences. Patients will only be included once
* Treatment with curative intent (surgery and/or (chemo)radio therapy)

Exclusion Criteria:

* Allergy to barium contrast
* Pregnancy or breastfeeding
* Inability or unwillingness to complete questionnaires and undergo examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Squamous cell carcinoma with any location in the oral cavity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified Barium Swallow Impairment profile (MBSImp) | Baseline, 2 and 12 months post-operative
  MBSImp is a 17-point assessment tool (0-55 points, a higher score indicates worse swallowing function) for interpreting MBSS that includes evaluation of the oral, pharyngeal and esophageal phase. The Penetration/Aspiration Scale will be applied for evaluating swallow safety ranging from 1 (no penetration/aspiration) to 8 (silent aspiration). The recordings as well as the interpretations are carried out by one of two trained otorhinolaryngologists.
MD Anderson Dysphagia Inventory (MDADI) | Baseline, 2 and 12 months post-operative
  The MDADI is a 20-item questionnaire assessing dysphagia-related QoL in head and neck cancer patients covering global, emotional, functional, and physical domains. The score ranges from 20 (poor function) to 100 (high function). The patient answers the questionnaire assisted by a nurse. A 10-point difference between groups in composite score is considered significant.
Days alive and out of hospital | 12 months post-operative
  During regular outpatient follow-up, the patient will be asked about hospital admission/re-admission since the last visit and the electronic chart will be accessed for verification of reason and length of stay.

SECONDARY OUTCOMES:
Weight | Baseline, 2 and 12 months post-operative
  Bodyweight will be measured at each visit
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) | Baseline, 2 and 12 months post-operative
  Scoring ranges from 0-100 where a high score in the functioning scales and global QoL indicate better functioning but for the symptom scales higher scores indicate higher symptom burden. The patient answers the questionnaires assisted by a nurse. A 10-point difference in instrument score is considered significant
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head And Neck 35 (EORTC H&N-35) | Baseline, 2 and 12 months post-operative
  Scoring ranges from 0-100 where a high score in the functioning scales and global QoL indicate better functioning but for the symptom scales higher scores indicate higher symptom burden. The patient answers the questionnaires assisted by a nurse. A 10-point difference in instrument score is considered significant
Functional oral intake score (FOIS) | Baseline, 2 and 12 months post-operative
  The patient will be asked about their food intake at each visit. FOIS is a 7 point scale regarding the level of oral intake, ranging from total tube dependency (1) to oral intake of a normal diet (7).

OTHER OUTCOMES:
Rehabilitation program | 12 months post-operatively
  At the 12-month follow-up a questionnaire will be sent to the patient's occupational therapist addressing the offered rehabilitation program (type and frequency). Patient satisfaction will be measured on a 10-point VAS-scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No